CLINICAL TRIAL: NCT06508216
Title: A Phase Ib/II, Open-label, Modular, Dose-finding and Dose-expansion Study to Explore Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of Novel Therapeutics in Patients With Early Relapsed Metastatic Triple-negative Breast Cancer
Brief Title: A Study to Explore Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of Novel Therapeutics in Patients With Early Relapsed Metastatic Triple-negative Breast Cancer
Acronym: COMPASS-TNBC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-503606-36-00; 2022/3571 (Other: CSET number)
Record Dates: First submitted 2024-07-03; First posted 2024-07-18 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: early relapsed metastatic; triple negative breast cancer; HER2 negative; Hormone-receptor negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: COMPASS-TNBC is a single-center, open-label, modular phase 1b/2 trial assessing the safety and efficacy of innovative therapies and combinations in patients with early relapsed advanced TNBC. The study is of modular design allowing assessment of safety, tolerability, and antitumor activity of multiple modules combining a wide range of different compounds. New combination treatment modules could be added during the study, via a protocol amendment. The combination module will be composed of 2 parts: a dose-finding part (Part 1) based on study drugs dose escalation and de-escalation and a dose-expansion part (Part 2) based on the RP2D found in Part 1. Modules for which the RP2D is already determined will be composed only of a dose-expansion part (Part 2). Therefore, the first 2 modules (Module 1: Dato-DXd single agent and Module 2: Dato-DXd + Durvalumab) will be composed only of part 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Module 1 of part 2 : Datopotamab Deruxtecan (Dato-DXd) Monotherapy (Experimental): Patients will receive Datopotamab Deruxtecan 6mg/kg every 21 days until progression or until unacceptable toxicity
  Interventions: Drug: Dato-DXd
- Module 2 of part 2 : Datopotamab Deruxtecan (Dato-DXd) + Durvalumab (Experimental): Patients will receive Datopotamab Deruxtecan 6mg/kg and durvalumab 1120mg every 21 days until progression or until unacceptable toxicity
  Interventions: Drug: Dato-DXd; Drug: Durvalumab

INTERVENTIONS:
Drug: Dato-DXd — Patients in module 1 & 2 will receive Datopotamab Deruxtecan (Dato-DXd) 6mg/kg every 21 days
Drug: Durvalumab — Patients in module 2 only will receive Durvalumab 1120mg every 21 days
  Arms: Module 2 of part 2 : Datopotamab Deruxtecan (Dato-DXd) + Durvalumab

SUMMARY:
Choice Of the Most Active Strategies for Short term recurring Triple Negative Breast Cancer:

A phase Ib/II, open-label, modular, dose-finding and dose-expansion study to explore safety, tolerability, pharmacokinetics, and anti-tumor activity of novel therapeutics in patients with early relapsed metastatic triple-negative breast cancer

DETAILED DESCRIPTION:
Every year, approximately 170.000 women are diagnosed with triple negative breast cancer (TNBC) and about 80-85% present with a stage II or III tumor making them eligible to neoadjuvant chemotherapy (NACT). Despite the substantial outcome improvements achieved with neoadjuvant chemotherapy-based strategies, at least 50-60% of patients with TNBC do not achieve pCR and are at higher risk of presenting with early disease recurrences. About 40% of patients with no-pCR experience distant recurrences within 12 months from the end of (neo)adjuvant treatments. Overall, 20-25% of patients with TNBC develop an early recurrence at ≤ 12 months from the end of (neo)adjuvant chemotherapy. Neither standard chemotherapy options nor approved targeted therapies exist for 35.000-40.000 women/year with TNBC (≈1200 women/year in France) that progress during (neo)adjuvant treatment or within 1 year from its termination. These patients present a "hard-to-treat" disease and a disproportionately high rate of morbidity and mortality. Notwithstanding, they are excluded from most current clinical trials that evaluate the efficacy of innovative strategies, with immunotherapy or targeting therapies in combination with chemotherapy. The treatment algorithm in 1st line is often based on the use of platine-containing regimens that provide very low response rates (less than 15%), no more than 2-3 months of 1st-line PFS and a median OS of about 9 months. Yet, comprehensive genomic analyses performed over the past years on patients with residual disease after neoadjuvant chemotherapy have not introduced concrete findings for guiding drug development in this setting. Comparisons of initial biopsies with post-NACT tumor tissues revealed a wide range of profound tumor changes acquired under the selective pressure of NACT that encompass the development of dominant subclones, tumor immune depletion and stem-cell phenotype enrichment that cannot be addressed with a single treatment strategy. Therefore, it is necessary to explore a broad range of treatment approaches to cover the different patterns involved. The idea is to set a rapidly recruiting phase I-II trials allowing to explore new treatment-strategies in patients with early recurrent and highly refractory TNBC have the potential to fulfil this utmost and urgent medical need.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients (who are ≥18 years of age at the time of signing the informed consent) who have a pathologically documented breast cancer that is:

   * Advanced/unresectable (patients who can be treated with curative intent are not eligible) or metastatic.
   * HER2-negative (IHC 0, 1+ or IHC 2+/ISH-) based on local assessment according to ASCO/CAP guidelines 1.
   * Documented as hormone receptor-negative (both oestrogen receptors and progesterone receptors are negative [oestrogen receptors and progesterone receptors < 10%]) as per GEFPICS guidelines in the metastatic setting 2.
2. Patients need to provide an adequate tissue sample: provided from either a new biopsy of a metastatic site or the most recent archival biopsy taken at the time of diagnosis of metastatic disease, if performed within 1 month of the ICF signature. Additionally, an archival sample of the primary tumor may be submitted (if available) in addition to any recent archival tissue provided.
3. Patients who have early relapsed triple negative breast cancer i.e.:

   * Patients who have received neo/adjuvant chemotherapy in the localized stage.
   * Radiological and anatomopathological evidence of disease recurrence or metastasis while on (neo)adjuvant treatment or within 12 months from the end of all treatments with curative intent.
4. Patients with germinal pathological BRCA1/2 mutations are eligible to the study if they have received prior treatment with PARP inhibitor.
5. ECOG PS of 0 to 2.
6. LVEF ≥ 50% within 28 days before enrolment.
7. Adequate organ and bone marrow function within 14 days prior to treatment assignment.
8. At least one lesion, not previously irradiated (and different from the biopsy site), that qualifies as a RECIST 1.1 target lesion at baseline.
9. An adequate treatment washout period before randomization/enrolment.
10. Patients with leptomeningeal or brain metastases can be included in the trial if symptoms are controlled with corticosteroids until 10 mg/day of prednisone or equivalent. Patients with brain metastases must receive radiotherapy if indicated, before study entry. Anticonvulsant therapy must be stable for at least 14 days prior to C1D1.

    Reproduction
11. Evidence of post-menopausal status or negative serum pregnancy test for females of child-bearing potential who are sexually active with a non-sterilized male partner.

    For women of child-bearing potential, a negative result for a pregnancy test (A negative serum pregnancy test at screening visit and a negative serum or urine pregnancy test within 72 hours prior to first study treatment administration).

    Women will be considered post-menopausal if they have been amenorrhoeic for at least 12 months without an alternative medical cause. The following age-specific requirements apply:
    * Women < 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.
    * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses> 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago).
12. Women who are surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) are eligible.
13. Female patients of child-bearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception from the time of screening and must agree to continue using such precautions for 7 months after the last dose of study treatment. Not all methods of contraception are highly effective. Female patients must refrain from egg cell donation and breastfeeding while on study and for 7 months after the last dose of study treatment. Not engaging in sexual activity for the duration of the study and drug washout period is an acceptable practice; however, periodic, or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.
14. Non-sterilized male patients who are sexually active with a female partner of child-bearing potential must use a condom with spermicide from screening to 4 months after the final dose of study treatment. Not engaging in sexual activity for the duration of the study and drug washout period is an acceptable practice; however, periodic, or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period. In addition, male patients should refrain from fathering a child or donating sperm during the study and for 4 months after the last dose of study treatment. Preservation of sperm should be considered prior to enrollment in this study.
15. Female patients must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study treatment administration. Preservation of ova should be considered prior to enrollment in this study Informed Consent
16. Patient must understand, sign and date the written informed consent form (ICF) prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedure as per protocol.
17. Patient must be affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

1. Evidence of untreated spinal cord compression or with leptomeningeal or brain metastases, requiring more than 10 mg/day of prednisone or equivalent.

   Note: Untreated spinal cord compression: patients can enter the study after adequate treatment of spinal cord compression.
2. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, uncontrolled or significant cardiovascular disease, severe pulmonary function compromise, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
3. Has a clinically significant corneal disease.
4. Has a history of non-infectious ILD/pneumonitis including radiation pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
5. Uncontrolled or significant lung disease or prior pneumonectomy.
6. Active connective tissue or inflammatory disorders requiring treatment, or active or prior documented autoimmune disease within the past 5 years. Of note, patients with vitiligo, Grave's disease or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. Patients with type 1 diabetes or hypothyroidism stable under treatment or not requiring systemic treatment are eligible.
7. Active primary immunodeficiency.
8. Has active or uncontrolled hepatitis B or C virus infection.

   Patients are eligible if they:
   1. Have been curatively treated for HCV infection as demonstrated clinically and by viral serologies
   2. Have received HBV vaccination with only anti-HBs positivity and no clinical signs of hepatitis
   3. Are HBsAg- and anti-HBc+ (i.e., those who have cleared HBV after infection) and meet conditions i-iii of criterion d below:
   4. Are HBsAg+ with chronic HBV infection (lasting 6 months or longer) and meet conditions i-iii below:

   i. HBV DNA viral load < 2000 IU/mL ii. Have normal transaminase values, or, if liver metastases are present, abnormal transaminases, with a result of AST/ALT <5× ULN, which are not attributable to HBV infection iii. Start or maintain antiviral treatment if clinically indicated as per the investigator
9. Patients with known controlled HIV infection and undetectable HIV-DNA are eligible to the trial.

   Note: all of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA, CD4+ count ≥ 350, no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti-HIV medications (meaning there are no expected further changes in that time to the number or type of antiretroviral drugs in the regimen). If an HIV infection meets the above criteria, monitoring of viral RNA load and CD4+ count is recommended. Patients must be tested for HIV during the screening period if acceptable by local regulations or an institutional review board (IRB)/ethics committee (EC).
10. Any concurrent systemic therapy (e.g. chemotherapy, targeted therapy, immunotherapy..), radiotherapy, investigational agent , or biological therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
11. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study treatment.
    2. Adequately treated non-melanoma skin cancer or Lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease.
12. Has a history of severe hypersensitivity reactions to either the study treatment(s) or inactive ingredients (including but not limited to polysorbate 80 of Dato-DXd), or has a history of severe hypersensitivity reactions to other monoclonal antibodies.
13. Patients having received prior treatment with any antibody drug conjugates targeting TROP2 (eg, Sacituzumab govitecan) are not eligible to the study.
14. Judgment by the Investigator that the patients should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
15. History of allogeneic organ transplantation.
16. Patient has clinically significant, uncontrolled heart disease and/or recent cardiac events including any of the following:

    1. History of angina pectoris, coronary artery bypass graft (CABG), symptomatic pericarditis, or myocardial infarction within 12 months prior to the start of study treatment.
    2. History of documented congestive heart failure (New York Heart Association functional classification III-IV).
    3. Documented cardiomyopathy.
    4. Patient has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO).
    5. History of any cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block), supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months.
    6. Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 100 mmHg, with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
17. Patients with prior use of immunosuppressive medications within 14 days prior to first study drug dose or anticipation of need for systemic immunosuppressive medication during study treatment, except for intranasal and inhaled corticosteroids or systemic corticosteroids at doses less than 10 mg/day of prednisone or equivalent.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 7 months after the last dose of study treatment. (See contraception requirements outlined in Appendix 7 of this protocol).
19. Administration of live attenuated vaccines within 30 days prior to the first dose of study treatment, or anticipation that such a live, attenuated vaccine will be required during the study or within 3 months after the last dose of study treatment.
20. Persons deprived of their freedom or under guardianship, or for whom it would be impossible to undergo the medical follow-up required by the trial, for geographic, social or psychological reasons.
21. Participation in another clinical study with an investigational product during the last 4 weeks prior to enrollment and while on study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Part 2_Efficacy of study therapies in each module_objective response rate (ORR) at 6 months. | Within the 6 months of treatment initiation
  ORR is defined as the proportion of patients who achieved a confirmed CR or PR within the 6 months of treatment initiation assessed by investigators.
Part 1_Safety and to determine the recommended phase II dose (RP2D) of study therapies in each module | During treatment_to be determined according to modules added later on
  measured by the DLTs, frequency and severity of any AEs, TEAEs, SAEs, AESIs graded according to NCI-CTCAE v5.0, proportion of treatment discontinuations, interruptions, and dose reductions due to any AEs; frequency and severity of laboratory abnormalities defined by NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Part 1&2_Progression free survival (PFS) | From the time date of the first dose until progression or death from any cause, whichever occurs first
  Defined as the time from the date of first dose until the date of the first objective documentation of disease progression or death from any cause, whichever occurs first. For patients without documented radiological progression, PFS will be censored at the date of last adequate radiological assessment without progression, unless death occurs within ≤ 2 missing assessments following the date of last known progression-free, in which case the death will be counted as a PFS event.
Part 1&2_Duration of response (DOR) | From cycle 3 (Week 6; each cycle is 28 days) up to 2 years after the EoT, an average of 33 months
  Defined as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progression (PD) or death due to any cause, whichever occurs first. Duration of response will be measured for responding patients (CR or PR) only.
Part 1&2_Clinical benefit rate (CBR) | During treatment period, a median of 6 months
  Defined as the proportion of patients with a complete (CR) or partial response (PR) or with stable disease (SD) > 6 months.
Part 1&2_Overall survival (OS) | From the date of the first dose until 24 months after EoT
  Defined as the time from the date of first dose until death. Patients alive at last follow-up will be censored at this date.
Part 2_Frequency of all adverse events | From enrollment to 30 days after EoT for module 1 and for 90 days for module 2
Part 2_Severity of all adverse events | From enrollment to 30 days after Eo for module 1 and for 90 days for module 2
  As defined by the NCI-CTCAE v5.0.
Part 2_Frequency of laboratory abnormalities | From enrollment until progression, median of 6 months
Severity of laboratory abnormalities | From enrollment until progression, median of 6 months
  Defined by NCI-CTCAE v5.0
Proportion of treatment discontinuation due to any AEs. | Treatment Period, median of 6 months
Proportion of treatment interruptions due to any AEs. | Treatment Period, median of 6 months
Proportion of dose reductions due to any AEs. | Treatment Period, median of 6 months
Part 1_efficacy of study therapies in each module_objective response rate (ORR) | Within the 6 months of treatment initiation
  ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) assessed by investigators. The objective response will be radiologically assessed every 6 weeks using RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pistillli, MD, Study Director — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, France